CLINICAL TRIAL: NCT01546740
Title: Glaucoma Prevalence in the Israeli Arab Population
Brief Title: Prevalence of Glaucoma in the Israeli Arab Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZIV-0060-11
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Glaucoma
Keywords: Glaucoma, Compliance, Prevalence
MeSH Terms: conditions — Glaucoma; Patient Compliance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glaucoma patients: all the ,medical records of patients who were diagnosed with primary open angle glaucoma, closed angle , pseudoexfoliative and neovascular glaucoma.

SUMMARY:
there is a variety of glaucoma prevalence within different populations. this study examine the prevalence of glaucoma in the Arab population in Israel' as well as the demographic variables and the compliance to treatment in the population.

DETAILED DESCRIPTION:
from Medical records of primary care clinic in the city of Tira. the patients are recruited, all glaucoma patients are above age of 20 years. they must suffer from CDR >= 0.5 with/without asymmetry with the other eye. or they suffer from glaucomatous damage to the visual fields.

ELIGIBILITY:
Inclusion Criteria:

* Cup-to-disk ratio (CDR) > 0.5 with asymmetry between the eyes
* Intraocular pressure (IOP) > 23 mm Hg
* Damage to the field of vision
* Age- above 20 Yrs. old

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinics from 1 Arab city in the center of Israel
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pikkel, M.D, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel